CLINICAL TRIAL: NCT04766827
Title: A Prospective Randomized Controlled Clinical Study of Albumin-bound Paclitaxel Combined With Cisplatin (AP Regimen) Versus Docetaxel Combined With Cisplatin (TP Regimen) Induced Chemotherapy in Advanced Head and Neck Squamous Tummor
Brief Title: Albumin-bound Paclitaxel Combined With Cisplatin Versus Docetaxel Combined With Cisplatin Induced Chemotherapy in Advanced Head and Neck Squamous Tummor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJCIHMF&ENT-001
Record Dates: First submitted 2021-01-29; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-11

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Albumin-Bound Paclitaxel; Docetaxel

STUDY DESIGN:
Intervention Model Description: A prospective randomized controlled clinical trail
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- albumin-bound paclitaxel combined with cisplatin (AP regimen) (Experimental): Paclitaxel (albumin combined type) 260 mg/m2, intravenous drip, d1, every three weeks for a cycle, a total of dosing 2 cycles; Cisplatin: 75 mg/m2, intravenous drip, d1, every three weeks for a cycle, a total of dosing 2 cycles;
  Interventions: Drug: albumin-bound paclitaxel
- docetaxel combined with cisplatin (TP regimen) (Active Comparator): docetaxel: 75 mg/m2, intravenous drip, d1, every three weeks for a cycle, a total of dosing 2 cycles; cisplatin: 75 mg/m2, d1 every three weeks for a cycle, a total of dosing 2 cycles;
  Interventions: Drug: albumin-bound paclitaxel

INTERVENTIONS:
Drug: albumin-bound paclitaxel — Paclitaxel for injection (albumin-bound) uses human serum albumin as the carrier to avoid the use of organic solvents for intravenous injection of paclitaxel, reducing the incidence of allergic reactions, and reducing the toxicity of the drug.
  Other Names: Docetaxel

SUMMARY:
Research Topic:

A prospective randomized controlled clinical study of albumin-bound paclitaxel combined with cisplatin (AP regimen) versus docetaxel combined with cisplatin (TP regimen) induced chemotherapy in advanced head and neck squamous cell carcinoma

Expected study duration:

Each subject received a 3-week regimen of AP or TP over 2 cycles.

Research objectives:

To evaluate the efficacy and safety of induction chemotherapy with albumin-bound paclitaxel in patients with advanced head and neck squamous cell carcinoma (HSCC), two induction chemotherapy regimens, AP regimen and TP regimen, were compared.

Trial Design. Single center, open label, controlled clinical study Number of cases: 116 Objective response rate (ORR=CR+PR) was used as the main evaluation index in this study.

DETAILED DESCRIPTION:
Research purposes:Research the effectiveness and safety of albumin-bound paclitaxel for induction chemotherapy in patients with advanced head and neck squamous cell carcinoma were evaluated,by comparing the AP regimen and the TP regimen .

Research content:To evaluate the effectiveness and safety of albumin-bound paclitaxel for induction chemotherapy in patients with advanced head and neck squamous cell carcinoma.

Study endpoint Primary endpoint: Objective response rate (ORR=CR+PR) (Assessed according to RECIST standards, see Annex 1) Secondary study endpoint: Surgical resection rate,Pathological remission rate,Progression-free survival (PFS), Overall survival (OS) Main safety indicators: Observe any adverse events that occurred in all subjects during the clinical study and within 1 month after stopping the drug, including clinical symptoms, abnormal vital signs, and abnormalities in laboratory examinations, and record their clinical features, Severity, time of occurrence, duration, treatment method and prognosis outcome, and determine its correlation with the study drug. The safety of the drug was evaluated according to the NCI-CTC AE 4.0 standard.

Study design:This is a single-center, open-label, controlled clinical study.The aime is observing and evaluating the effectiveness and safety of albumin-bound paclitaxel for induction chemotherapy in patients with advanced head and neck squamous cell carcinoma.

This study is planned to be carried out in Tianjin Cancer Hospital. According to the research principles of GCP.

The study plans to recruit 116 qualified subjects. This study used objective response rate (ORR=CR+PR) as the main evaluation index. According to previous reports, the ORR of the TP group was 50%, and the ORR of the AP group was estimated to be 75%. The test level is set to 0.05 on one side, the test power is set to 0.8, and the estimated dropout rate is 20%. Using the Logrank-Lakatos algorithm, the total sample size is calculated to be 116 cases.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Age ≥18 years old, male or female;
  2. Subjects had squamous cell carcinoma of the head and neck confirmed by histrohistology or cytology;
  3. CLINICAL STAGE III OR IV WITHOUT DISTANT METASTASES (AJCC 8th)
  4. Patients who have not previously received initial treatment with chemotherapy or radiation;
  5. KPS acuity 70;
  6. Normal bone marrow reserve function and normal liver and kidney function;
  7. Expected survival time ≥3 months;
  8. Subjects of child-bearing age must agree to use effective contraceptive measures during the study period; The serum or urine pregnancy test must be negative for women of childbearing age 72 hours before the start of chemotherapy;
  9. Subjects have good compliance, can carry out treatment and follow-up, and voluntarily abide by the regulations of this study;
  10. Subjects voluntarily sign the informed consent.

Exclusion Criteria:

* Exclusion criteria:

  1. Patients with distant metastasis;
  2. The presence of uncontrolled serious medical diseases, such as combined with serious medical diseases, including serious heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.;
  3. The presence of dementia, altered mental status or any mental illness that would prevent understanding or giving informed consent or filling out questionnaires;
  4. Subjects with grade ≥2 peripheral neuropathy according to CTCAE V5.0;
  5. A history of allergy or hypersensitivity to any therapeutic ingredient;
  6. Suffered from malignant tumors other than squamous cell carcinoma of the head and neck in the past 5 years, except adequately treated basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery;
  7. Abnormal results of physical and laboratory tests:

     A) Hematologic abnormalities are defined as:

     I) Absolute count of neutrophils (ANC) : < 1.5×109 / L; Ii) Platelet (PLT) count: < 100×109/L; Iii) Hemoglobin (Hb) level < 90g/L;

     B) Abnormal liver function is defined as:

     I) Total bilirubin (TBIL) level: 1.5 times of the upper limit of normal value of > (ULN); Ii) AST and ALT levels of >ULN were 2.5 times, and BBB>N was 5 times if liver metastasis was present;

     C) Definition of abnormal renal function:

     1.5 times of serum creatinine > ULN, or the calculated creatinine clearance rate < 50ml/min;
  8. Patients who need to be treated with other anti-tumor drugs;
  9. Has received any other investigational drug therapy or participated in another interventional clinical trial within 30 days prior to screening;
  10. The researcher considers it unsuitable for inclusion;
  11. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 21 days
  ORR=CR+PR

SECONDARY OUTCOMES:
Surgical resection rate | 1 month
  the rate of Surgical resection in all samples
pathological response rate | 1 month
  the rate of pathological response in all samples
PFS | 5 year
  progression-free survival
OS | 5 year
  overall survival

OTHER OUTCOMES:
Incidence of adverse events | 90 days
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xudong Wang, MD, Principal Investigator — Tianjin Medical University Cancer Institute & Hospital, National Clinical Research Center of Cancer
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China